CLINICAL TRIAL: NCT04571775
Title: Investigation of Possible Effects of a Lifestyle Product in a Double-blind Pre-Post-Between-Groups Study
Brief Title: Effects of a Lifestyle Product on Physiological Measures and Subjective Well-being in Humans: A Systematic Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Waveguard GmbH (Industry)
Collaborators: University of Stuttgart, Institute of Human Factors and Technology Management (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: WAVEGUARD STRESS HUMANS FR01
Record Dates: First submitted 2020-09-14; First posted 2020-10-01 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2020-09

CONDITIONS: Healthy Lifestyle
Keywords: EEG; ECG; EDA; resting state; well-being; stress; sleep

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Qi-Shield user group (Active Comparator)
  Interventions: Device: Qi-Shield user group
- Sham Qi-Shield user group (Sham Comparator)
  Interventions: Device: Sham Qi-Shield user group
- No Qi-Shield device group (No Intervention)

INTERVENTIONS:
Device: Qi-Shield user group — real device Qi-Shield (treatment)
  Arms: Qi-Shield user group
Device: Sham Qi-Shield user group — sham device (placebo)
  Arms: Sham Qi-Shield user group

SUMMARY:
Research question: The study investigates possible effects of the lifestyle product "Qi-Shield" on a subjective and (neuro-)physiological level. Thereby, effects on well-being, stress perception and the sleep quality as well as influencing factors like personality and beliefs are of particular interest.

Sample and Design: In the study 90 test persons are to be tested in a double-blind pre-post between-subject design with three groups (real device (A) - sham device without effectiveness (also called placebo, B) - no device (C)).

Measurement methods: Established questionnaires and scales as well as (neuro-)physiological methods comprising electroencephalography (EEG), electrocardiogram (ECG) and skin conductance level measure (electrodermal activity, EDA) during a 20 mins resting state measure with alternating eyes open and closed are used.

Statistical evaluation: Group comparisons (A, B, C) in the difference between the measurement points (post - pre) on a subjective and (neuro-)physiological level.

DETAILED DESCRIPTION:
Within this study, the Lifestyle product Qi-Shield manufactured by Waveguard GmbH shall be investigated regarding its subjective psychological and neurophysiological effects. Thereby, the constructs well-being, stress feeling in the everyday life and subjectively perceived sleep quality as well as (neuro)-physiological correlates are of particular interest. The physical effects of the product will not be scope of this study. According to the World Health Organization (WHO), the number and variety of sources of electromagnetic fields (EMF) has increased over the last decades. These sources include video display units (VDUs) associated with computers, cell phones and their base stations, which does not exclude possible health risks from EMF emissions. In this context, several studies report a variety of health problems associated with exposure to EMFs. The sensitivity to EMF is called electromagnetic hypersensitivity. EHS is characterized by a variety of non-specific effects that people attribute to exposure to EMFs. Among the most frequently reported effects are dermatological symptoms and neurasthenic and vegetative symptoms. Some laboratory studies explored the relationship between EMF (short-term exposure) and EHS and observed highly inter-subjectively varying effects. However, EHS has no clear diagnostic criteria and there is no scientific basis to link EHS effects to EMF exposure, at least not to short-term EMF exposure. However, the limited quantity and quality of research on possible effects of EMF does not allow excluding long-term effects.

The Qi-Shield device aims to reduce effects of EMF exposure and enable to maintain subjective well-being, low stress perception and good sleep quality.

Previous literature reported neuronal correlates characterized with (acute) stress exposure and effects on well-being (especially emotional regulation) at the physiological (autonomic nervous system) and neurophysiological level (central nervous system). These measurements can also be observed during the resting state. On a physiological level, heart rate variability (HRV) -recorded by the electrocardiography (ECG) - can be derived as a constant measure of the influence of stress. The most frequently reported parameter under acute stress was low parasympathetic activity, characterized by a decrease in the high frequency band (0.15-0.4 Hz, HF) and an increase in the low frequency band (0.04-0.15 Hz, LF). Furthermore, the measurement of sweat production of the skin - recorded by the derivation of the electrodermal skin activity (EDA) - is suitable to characterize specific influences on the autonomic nervous system. For this purpose, the EDA signal can be segmented into phasic reactions (individual rapid reactions - usually responses to a given stimulus) and tonic components (longer lasting basic skin resistance value). From these two components, the number of individual phasic responses, the summed amplitude of the phasic responses, and the change in the tonic state of the electrical conductivity are the most suitable feature to investigate effects of stress on the physiological level. On a neurophysiological level, acute stress leads to effects in the resting state networks of the brain. A recently published study showed that acute stress weakens the connectivity of the front-parietal module and strengthens the connectivity of the module in the default mode network. Thus, it can be assumed that stress influences the information flow in networks that are important for salience processing (especially attention control) and self-referential mental processing or even emotional processing. Possible quantitative markers from EEG resting state measurements are the derivation of the frequency spectrum (derived by calculating the Fourier transform) as well as connectivity measures (calculating coherence measures from the EEG frequency spectrum). In particular, the ratio of frontal theta (4-7 Hz) to beta (13-30 Hz) activity can be derived from the resting EEG as an indicator of possible influences on cognitive control abilities (attention-control). Possible influences on one's own well-being, such as the ability to control one's emotions (impulse control), can be observed in changes in frontal alpha (8-14 Hz) activity both in frequency spectrum and coherence and in the determination of so-called frontal alpha asymmetry. Since there could be possible effects of Qi-shield may result in a reduction of EMF, power and coherence measures in individual alpha and beta band resting activity already observed in connection with EMF exposure may serve as a basis for this study. Regarding subjective influences on effects of the here studied device, various studies reported correlations between personality characteristics (i.e, critical thinking), fluid intelligence and the tendency towards and openness for paranormal beliefs. Matrix intelligence tests such as the Vienna Matrix Test 2 (WMT-2) detect inferential thinking and correlate strongly positively with manifestations in critical thinking. Both constructs show a negative correlation between manifestations of paranormal beliefs and statements about paranormal experiences. An influence of personality factors such as openness to new experiences can also be assumed. To control possible moderating or mediating factors, these constructs will be investigate, too.

The study design is a double-blind Pre-Post Between-Subject Design. This means that the subjects are invited twice (pre-session and post-session). Between the two sessions, there is one week of exposure time during which the subjects of the invention groups take the device home.

At the beginning of the experiment in the pre-session, all subjects (N=90) are checked for the presence of inclusion and exclusion criteria and if necessary excluded from the study. The subjects are assigned to the trial groups in a semi-randomized latin-square counterbalanced manner. The assignment is double-blind, i.e. neither the volunteer nor the investigator is informed which group receives a placebo or real intervention. The real devices resemble the sham devices in appearance, composition and weight, so that a traceability based on these factors is not possible. The products are marked with the letters A and B. The assignment which letter belongs to which intervention group is explained in a sealed envelope and will be opened after completion of the study and analysis. Prior to the start of the study, participants are informed about their rights and potential risk of participation with an authorized deception in case of the assumed effects of the intervention and asked to sign the declaration of consent in line with the declaration of Helsinki. The information for the intervention groups differs from the information for the no-intervention group, as the latter serves as a control group and therefore does not receive any information about the intervention.

Afterwards the test person is asked to answer a control item for the examined product (only for group A - correct product and B - sham product) and then fill in questionnaires about sleep quality and current fatigue (in detail below). Subsequently, the sensors for EEG, ECG and EDA are prepared and fixed to the head and body accordance with the corresponding guidelines. After this preparation, the resting state measurements of electrophysiological signals (EEG, ECG and EDA) are recorded during relaxation. In order to identify possible effects in the alpha band, resting measurements are taken with eyes closed (so-called eyes closed EC) as well as with eyes open (so-called eyes open, EO) according to a standardized procedure. This consists of an alternating task (20 minutes in total) in which the subjects are asked to alternately "relax with eyes open" and "relax with eyes closed" for 60 seconds each. In the phase with open eyes, the test persons are asked to fixate a crosshair on a screen. The change between the phases is signalled by an acoustic tone.

Afterwards, the measurement equipment is removed from the head and body and the test person is asked to answer several questionnaires and scales (in detail below).

At the end of the session, test persons from groups A and B receive the information on handling the device and the device with the respective label (A or B). During the seven days exposure period, subjects are asked daily to answer questions about their current condition and special events via an online survey. The subjects in groups A and B are also asked to answer two questions related to the handling of the product. During the exposure period, subjects are supervised via WhatsApp or E-mail from employees of the University of Stuttgart and Fraunhofer IAO. A short standardized text will be used as a reminder to fill in the questionnaires if participants have not been completed by a certain time (6 pm). The second session is similar to the first session in terms of the way the study is conducted. At the beginning of the session, the subjects are again given detailed written information about the study and asked to sign the declaration of consent for the second session. Afterwards the participants are asked to fill in the daily questions about well-being, everyday stress and special events as well as the questionnaires about sleep quality and current fatigue. Afterwards, we will conduct the neurophysiological measurement during the resting state as in the pre-session. Afterwards, the measurement sensors are removed from the head and body and the participant is asked to answer the questionnaires and scales. At the end of the post-session the test persons will be informed in detailed and the deception will be dissolved. The experimenter will answers further questions.

ELIGIBILITY:
Inclusion Criteria:

* healthy males and females (approximately 50:50)
* sufficient language skills
* No knowledge or experience with the Qi-Shield device

Exclusion Criteria:

* neurological diseases such as e.g. epilepsy or psychiatric disorders (asked for by selfdisclosure) or the intake of centrally effective drugs, as these factors can influence electrophysiological signals such as EEG ECG and EDA.
* persons with COVID risk factors

Since it has been repeatedly reported that EHS individuals are prone to certain physiological reactions that are outside the normal range, we will exclude these individuals in the present study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-10-03 (Actual); Primary Completion 2021-02-01 (Estimated); Study Completion 2021-02-01 (Estimated)

PRIMARY OUTCOMES:
Adapted Pittsburgh Sleep Quality Index (PSQI) | Change from Baseline Measure at the 1st day at 7 days
  The PSQI asks about sleep quality retrospectively. It asks about the frequency of sleep disturbing events, the estimation of sleep quality, the usual sleeping times, sleep latency and sleep duration, the intake of sleep medication, as well as daytime tiredness. A total of 18 items are used for quantitative evaluation and 7 components are assigned, each of which can assume a value range from 0 to 3. The total score results from the summation of the component scores and can vary from 0 to 21, whereby a higher value corresponds to a reduced sleep quality. There is an empirically determined cut-off value (from 5), which allows a division into "good" and "bad" sleepers. Lower values are associated with better sleep quality.
WHO-5 | Change from Baseline Measure at the 1st day at 7 days
  The WHO 5 Well-being Index is a short questionnaire of only five questions that measures well-being. Values from 0 to 5 can be entered for each question. By summing up the values for the answers, one obtains a total value, whereby a low total value corresponds to a low level of well-being. A value less than 13 should indicate a possible depression. Standard values and test quality criteria can be used for WHO-5. The processing time is less than one minute.
State Trait Anxiety Inventory | Change from Baseline Measure at the 1st day at 7 days
  The State Trait Anxiety Inventory is based on the distinction between anxiety as a state and anxiety as a characteristic. The two scales of the STAI, each with 20 items, serve to record fear as a state (state anxiety) and fear as a characteristic (trait anxiety). The answer format is a 4-point Likert-rating scale. Higher values indicate higher state or trait anxiety.
Positive and Negative Affect Schedule , PANAS | Change from Baseline Measure at the 1st day at 7 days
  The PANAS records the emotional state of mind. The questionnaire consists of 20 adjectives that describe different sensations and feelings. 20 adjectives describe the dimensions of positive (10) and negative affect (10). The PANAS is used in this study for two temporal dimensions - once for an immediate assessment and further for a period of one week. The answer format is a 5-point Likert-rating scale (1 = "not at all" and 5 = " extremely").
Adapted Perceived Stress Scale | Change from Baseline Measure at the 1st day at 7 days
  The scale of perceived stress asks for subjectively experienced stress retrospectively. The 10 items were validated on a German sample and are a reliable, valid and economic instrument for the assessment of perceived stress. The answer format is a 7-point Likert-rating scale (1 = " not at all" and 7 = "completely"). Higher values are related to more stress perception.
Brief Resilience Scale | Change from Baseline Measure at the 1st day at 7 days
  The Brief Resilience Scale is a short, six-item measure of the ability to recover from stress on a five-point Likert scale. It showed good psychometric characteristics with high internal consistency and reliability in repeat tests.The items are rated on a five-point Likert scale (1 = strongly disagree, 2 = disagree, 3 = neutral, 4 = agree, 5 = strongly agree or 1 = stimme überhaupt nicht zu, 2 = stimme eher nicht zu, 3 = neutral, 4 = stimme eher zu, 5 = stimme vollkommen zu, respectively). A higher score is associated with a higher ability to cope stressfull events and higher stress resilience.
EEG Alpha band power | Change from Baseline Measure at the 1st day at 7 days
EEG Alpha band functional connectivity | Change from Baseline Measure at the 1st day at 7 days
EEG Beta band power | Change from Baseline Measure at the 1st day at 7 days
EEG Beta band functional connectivity | Change from Baseline Measure at the 1st day at 7 days
EEG: Frontal alpha band asymmetry (right side activity) | Change from Baseline Measure at the 1st day at 7 days
EEG: Frontal theta/beta band ratio | Change from Baseline Measure at the 1st day at 7 days
EDA: number of individual phasic responses | Change from Baseline Measure at the 1st day at 7 days
EDA: number of summed amplitude of phasic responses | Change from Baseline Measure at the 1st day at 7 days
ECG: Low frequency response in the heart rate variability | Change from Baseline Measure at the 1st day at 7 days
ECG: High frequency response in the heart rate variability | Change from Baseline Measure at the 1st day at 7 days
ECG: Average heart rate | Change from Baseline Measure at the 1st day at 7 days
ECG: Standard deviation of normal to normal intervals (SDNN) | Change from Baseline Measure at the 1st day at 7 days
Satisfaction with Life Scale | Change from Baseline Measure at the 1st day at 7 days
  The five-item scale is used to measure life satisfaction. This is understood as a multifactorial construct with affective and cognitive-evaluative components. The affective components are characterized by the presence of positive and the absence of negative emotions. The cognitive-evaluative components are composed of global and domain-specific satisfaction in different areas of life. The response format is a 7-point Likert-rating scale (1 = "not at all" and 7 = "completely").

SECONDARY OUTCOMES:
Complementary and Alternative Medicine (CAM) Health Belief Questionnaire | Change from Baseline Measure at the 1st day at 7 days
  The questionnaire collects the attitude and openness towards complementary and alternative medicine. It uses 10 items with a 7-point Likert-rating scale (1 = "not at all" and 7 = "completely"). Higher values are related to stronger beliefs in complementary and alternative medicines (CAM).
Adapted Paranormal Experience Scale | Change from Baseline Measure at the 1st day at 7 days
  The adapted scale for paranormal experiences asks in 12 items experiences of supernatural phenomena with a binary answer format. Higher values are related to stronger beliefs in and susceptibility for paranormal experiences.
Revised Paranormal Belief Scale | Change from Baseline Measure at the 1st day at 7 days
  With 26 items, the scale of paranormal beliefs in the seven dimensions of Traditional Religious Belief, Psi, Witchcraft, Superstition, Spiritualism, Extraordinary Life Forms and Precognition asks. A 7-point Likert rating scale is used as the answer format (1 = "not at all" and 7 = " completely"). Higher values are related to stronger susceptibility for paranormal beliefs.
Vienna matrix test | 1st day [Pre-session]
  The WMT-2 is a shortened version of the Vienna Matrices Test with rapidly scaled 18 items. Depending on the type of item, the test measures the ability to reason when dealing with abstract symbols. According to Cattell, this can be classified as fluid intelligence (ability to think logically, recognize connections and figural relationships and find solutions to problems), which is largely independent of learning experience and culture. The concept of the WMT is based on that of Raven's Progressive Matrices. Higher values indicate higher ability in fluid intelligence.
Short version of the Big 5 Inventory | 1st day [Pre-session]
  The short version of the Big 5 inventory includes the personality dimensions openness to experience, conscientiousness, extraversion, tolerance and neuroticism. The inventory uses 21 items with a 7-point likert scale (1 -strongly disagress to 7 strongly agree) and is considered economic with an average processing time of less than 2 minutes. The results show satisfactory psychometric parameters for the BFI-K. In addition to sufficient reliability, the factorial validity of the procedure as well as high agreement with acquaintance judgements and with other established procedures for recording the five-factor model could be confirmed.
Karolinska Sleepiness Scale | Change from Baseline Measure at the 1st day at 7 days
  The Karolinska Sleepiness Scale asks for the currently felt fatigue in an item on a scale from 0 to 9. The scale can also be displayed via a visual analogue scale. High values are correlates with high sleepiness.

CONTACTS AND LOCATIONS:
Overall Officials: Katharina Lingelbach, Principal Investigator — Fraunhofer Institute for Industrial Engineering IAO
Locations (1):
- Fraunhofer Institute for Industrial Engineering IAO, Stuttgart, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akerstedt T, Gillberg M. Subjective and objective sleepiness in the active individual. Int J Neurosci. 1990 May;52(1-2):29-37. doi: 10.3109/00207459008994241. PMID 2265922
- [Background] Angelidis A, van der Does W, Schakel L, Putman P. Frontal EEG theta/beta ratio as an electrophysiological marker for attentional control and its test-retest reliability. Biol Psychol. 2016 Dec;121(Pt A):49-52. doi: 10.1016/j.biopsycho.2016.09.008. Epub 2016 Sep 30. PMID 27697551
- [Background] Aubeck, H.-J. (1989). Querschnitt der Parapsychologie. Eine Einführung in die okkulte Wissenschaft. Deutschland, Frankfurt a. M.: R. G. Fischer.
- [Background] Augner C, Gnambs T, Winker R, Barth A. Acute effects of electromagnetic fields emitted by GSM mobile phones on subjective well-being and physiological reactions: a meta-analysis. Sci Total Environ. 2012 May 1;424:11-5. doi: 10.1016/j.scitotenv.2012.02.034. Epub 2012 Mar 14. PMID 22421088
- [Background] Blankertz, B., Sanelli, C., Halder, S., Hammer, E., Kübler, A., Müller, K. R., ... & Dickhaus, T. (2009). Predicting BCI performance to study BCI illiteracy. BMC Neuroscience, 10(Suppl 1), 84. doi: 10.1016/j.neuroimage.2010.03.022
- [Background] Bortz, J., & Döring, N. (2006). Forschungsmethoden und Evaluation: für Human- und Sozialwissenschaftler. Heidelberg, de: Springer-Medizin-Verl.
- [Background] Breyer, B., & Bluemke, M. (2016). Deutsche Version der Positive and Negative Affect Schedule PANAS (GESIS Panel). Zusammenstellung sozialwissenschaftlicher Items und Skalen (ZIS). https://doi.org/10.6102/zis242
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Chmitorz A, Wenzel M, Stieglitz RD, Kunzler A, Bagusat C, Helmreich I, Gerlicher A, Kampa M, Kubiak T, Kalisch R, Lieb K, Tuscher O. Population-based validation of a German version of the Brief Resilience Scale. PLoS One. 2018 Feb 13;13(2):e0192761. doi: 10.1371/journal.pone.0192761. eCollection 2018. PMID 29438435
- [Background] Danker-Hopfe H, Eggert T, Dorn H, Sauter C. Effects of RF-EMF on the Human Resting-State EEG-the Inconsistencies in the Consistency. Part 1: Non-Exposure-Related Limitations of Comparability Between Studies. Bioelectromagnetics. 2019 Jul;40(5):291-318. doi: 10.1002/bem.22194. Epub 2019 Jun 18. PMID 31215052
- [Background] Dishman RK, Nakamura Y, Garcia ME, Thompson RW, Dunn AL, Blair SN. Heart rate variability, trait anxiety, and perceived stress among physically fit men and women. Int J Psychophysiol. 2000 Aug;37(2):121-33. doi: 10.1016/s0167-8760(00)00085-4. PMID 10831999
- [Background] Eid, M., Gollwitzer, M., & Schmitt, M. (2017). Statistik und Forschungsmethoden: mit Online-Materialien. Weinheim, Basel, de: Beltz Verlag.
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Formann, A. K., & Piswanger, K. (1979). WMT-2. Wiener Matrizen-Test. Ein Rasch-skalierter sprachfreier Intelligenztest. Göttingen: Hofgrefe Testzentrale.
- [Background] Hergovich, A. (2003). Field dependence, suggestibility and belief in paranormal phenomena. Personality and Individual Differences, 34, 195-209. https://doi.org/10.1016/S0191-8869(02)00022-3
- [Background] Hergovich, A., & Arendasy, M. (2005). Critical thinking ability and belief in the paranormal. Personality and Individual Differences, 38, 1805-1812. https://doi.org/10.1016/j.paid.2004.11.008
- [Background] Imperatori C, Farina B, Valenti EM, Di Poce A, D'Ari S, De Rossi E, Murgia C, Carbone GA, Massullo C, Della Marca G. Is resting state frontal alpha connectivity asymmetry a useful index to assess depressive symptoms? A preliminary investigation in a sample of university students. J Affect Disord. 2019 Oct 1;257:152-159. doi: 10.1016/j.jad.2019.07.034. Epub 2019 Jul 5. PMID 31301617
- [Background] Janke, S., & Glöckner-Rist, A. (2012). Deutsche Version der Satisfaction with Life Scale (SWLS). Zusammenstellung sozialwissenschaftlicher Items und Skalen (ZIS). https://doi.org/10.6102/zis147
- [Background] Kim HG, Cheon EJ, Bai DS, Lee YH, Koo BH. Stress and Heart Rate Variability: A Meta-Analysis and Review of the Literature. Psychiatry Investig. 2018 Mar;15(3):235-245. doi: 10.30773/pi.2017.08.17. Epub 2018 Feb 28. PMID 29486547
- [Background] Laux, L., Glanzmann, P., Schaffner, P., & Spielberger, C. D. (1981). Das State-Trait-Angstinventar (STAI). Weinheim, DE: Beltz.
- [Background] Lie D, Boker J. Development and validation of the CAM Health Belief Questionnaire (CHBQ) and CAM use and attitudes amongst medical students. BMC Med Educ. 2004 Jan 12;4:2. doi: 10.1186/1472-6920-4-2. PMID 14718061
- [Background] Psychiatric Research Unit, WHO Collaborating Center for Mental Health, WHO-5 Frederiksborg General Hospital, DK-3400 Hillerød. Abgerufen am 01.07.2020 unter https://www.thieme.de/de/thieme-telecare/143343.htm
- [Background] Rammstedt, B., & John, O. P. (2005). Kurzversion des big five inventory (BFI-K). Diagnostica, 51, 195-206.
- [Background] Rubin GJ, Das Munshi J, Wessely S. Electromagnetic hypersensitivity: a systematic review of provocation studies. Psychosom Med. 2005 Mar-Apr;67(2):224-32. doi: 10.1097/01.psy.0000155664.13300.64. PMID 15784787
- [Background] Seitz H, Stinner D, Eikmann T, Herr C, Roosli M. Electromagnetic hypersensitivity (EHS) and subjective health complaints associated with electromagnetic fields of mobile phone communication--a literature review published between 2000 and 2004. Sci Total Environ. 2005 Oct 15;349(1-3):45-55. doi: 10.1016/j.scitotenv.2005.05.009. Epub 2005 Jun 21. PMID 15975631
- [Background] Schneider EE, Schonfelder S, Domke-Wolf M, Wessa M. Measuring stress in clinical and nonclinical subjects using a German adaptation of the Perceived Stress Scale. Int J Clin Health Psychol. 2020 May-Aug;20(2):173-181. doi: 10.1016/j.ijchp.2020.03.004. Epub 2020 May 22. PMID 32550857
- [Background] Shen HH. Core Concept: Resting-state connectivity. Proc Natl Acad Sci U S A. 2015 Nov 17;112(46):14115-6. doi: 10.1073/pnas.1518785112. No abstract available. PMID 26578753
- [Background] van Son D, de Rover M, De Blasio FM, van der Does W, Barry RJ, Putman P. Electroencephalography theta/beta ratio covaries with mind wandering and functional connectivity in the executive control network. Ann N Y Acad Sci. 2019 Sep;1452(1):52-64. doi: 10.1111/nyas.14180. Epub 2019 Jul 16. PMID 31310007
- [Background] Tobacyk, J. (2004). A Revised Paranomal Belief Scale. International Journal of Transpersonal Studies, 23, 94 - 98. doi:10.1037/t14015-000
- [Background] Wallace J, Selmaoui B. Effect of mobile phone radiofrequency signal on the alpha rhythm of human waking EEG: A review. Environ Res. 2019 Aug;175:274-286. doi: 10.1016/j.envres.2019.05.016. Epub 2019 May 12. PMID 31146099
- [Background] Watson G., & Glaser E.M., (1991). Watson-Glaser Critical Thinking Appraisal Manual. London: Psychological Corporation
- [Background] WHO (2004, October 25 -27). WHO workshop on electromagnetic hypersensitivity. Prague, Czech Republic. Abgerufen am 01.07.2020 unter https://www.who.int/peh-emf/meetings/hypersensitivity_prague2004/en/
- [Background] Zhang Y, Dai Z, Hu J, Qin S, Yu R, Sun Y. Stress-induced changes in modular organizations of human brain functional networks. Neurobiol Stress. 2020 May 25;13:100231. doi: 10.1016/j.ynstr.2020.100231. eCollection 2020 Nov. PMID 32490057
- [Background] Zhang, J., Hua, Y., Xiu, L., Oei, T. P., & Hu, P. (2020). Resting state frontal alpha asymmetry predicts emotion regulation difficulties in impulse control. Personality and Individual Differences, 159, 109870. https://doi.org/10.1016/j.paid.2020.109870
- [Background] Nolte G, Bai O, Wheaton L, Mari Z, Vorbach S, Hallett M. Identifying true brain interaction from EEG data using the imaginary part of coherency. Clin Neurophysiol. 2004 Oct;115(10):2292-307. doi: 10.1016/j.clinph.2004.04.029. PMID 15351371
- [Background] Ewald A, Marzetti L, Zappasodi F, Meinecke FC, Nolte G. Estimating true brain connectivity from EEG/MEG data invariant to linear and static transformations in sensor space. Neuroimage. 2012 Mar;60(1):476-88. doi: 10.1016/j.neuroimage.2011.11.084. Epub 2011 Dec 7. PMID 22178298
- [Background] Lachaux JP, Rodriguez E, Martinerie J, Varela FJ. Measuring phase synchrony in brain signals. Hum Brain Mapp. 1999;8(4):194-208. doi: 10.1002/(sici)1097-0193(1999)8:43.0.co;2-c. PMID 10619414
- [Background] Bruna R, Maestu F, Pereda E. Phase locking value revisited: teaching new tricks to an old dog. J Neural Eng. 2018 Oct;15(5):056011. doi: 10.1088/1741-2552/aacfe4. Epub 2018 Jun 28. PMID 29952757
- [Background] Stam CJ, Nolte G, Daffertshofer A. Phase lag index: assessment of functional connectivity from multi channel EEG and MEG with diminished bias from common sources. Hum Brain Mapp. 2007 Nov;28(11):1178-93. doi: 10.1002/hbm.20346. PMID 17266107
- [Background] Vinck M, Oostenveld R, van Wingerden M, Battaglia F, Pennartz CM. An improved index of phase-synchronization for electrophysiological data in the presence of volume-conduction, noise and sample-size bias. Neuroimage. 2011 Apr 15;55(4):1548-65. doi: 10.1016/j.neuroimage.2011.01.055. Epub 2011 Jan 27. PMID 21276857
- [Background] Pan J, Tompkins WJ. A real-time QRS detection algorithm. IEEE Trans Biomed Eng. 1985 Mar;32(3):230-6. doi: 10.1109/TBME.1985.325532. No abstract available. PMID 3997178

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-09-20): https://cdn.clinicaltrials.gov/large-docs/75/NCT04571775/Prot_SAP_000.pdf
  • Informed Consent Form (2020-09-20): https://cdn.clinicaltrials.gov/large-docs/75/NCT04571775/ICF_001.pdf